CLINICAL TRIAL: NCT07007520
Title: An Open-label, Randomized, Single-dose, Crossover Study to Evaluate the Food Effect on the Pharmacokinetics of DA-5223 in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Food Effect on the Pharmacokinetics of DA-5223 in Healthy Adult Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: DA5223_FE_I
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Healthy Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental)
  Interventions: Drug: DA-5223(Fasting); Drug: DA-5223(Fed)
- Sequence B (Experimental)
  Interventions: Drug: DA-5223(Fasting); Drug: DA-5223(Fed)

INTERVENTIONS:
Drug: DA-5223(Fasting) — once a day
Drug: DA-5223(Fed) — once a day

SUMMARY:
This study will evaluate the food effect on the pharmacokinetics of DA-5223 in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female, 19 years to 55 years
* Male weighing 50 kg or more, female weighing 45 kg or more with a body mass index (BMI) of 18.0 kg/m2 to 30.0 kg/m2
* The subjects signed and dated informed consent form after hearing a detailed explanation of the study, fully understanding and determined voluntarily to participate

Exclusion Criteria:

* The subjects with acute illness
* The subjects with a history of gastrointestinal disease or surgery that may affect the absorption of Investigational Product
* The subjects hypersensitive to any of the Investigational Product components or other drug components
* The subjects who have continuously consumed excessive smoking or alcohol within 6 months of screening, or who cannot stop smoking, caffeine, or alcohol intake during hospitalization
* The subjects who are pregnant or lactating

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
AUC-last | 0~12 hours
  Area under the plasma concentration-time curve up to the last measurable concentration
Cmax | 0~12 hours
  Peak Plasma Concentration

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Global Clinical Trials Center, Seongnam-si, Gyeonggi-do, South Korea